CLINICAL TRIAL: NCT01406431
Title: A Single Dose, Sequence-randomized, Open-label, 2x2 Crossover Study to Compare Pharmacokinetics Between Pitavastatin and Valsartan Co-administration and Livalo® Fixed Combination Drug in Healthy Male Subjects
Brief Title: Pharmacokinetic Study of Livalo® Fixed Combination Drug in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: JW-PTV-102
Record Dates: First submitted 2011-07-26; First posted 2011-08-01 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Hyperlipidemia; Hypertension
Keywords: pitavastatin; Livalo
MeSH Terms: conditions — Hyperlipidemias; Hypertension | interventions — pitavastatin; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitavastatin + Valsartan (Active Comparator): Intervention: Drug: Pitavastatin, Valsartan
  Interventions: Drug: Pitavastatin, Valsartan
- Livalo fixed combination drug (Experimental): Intervention: Drug: Livalo® fixed combination drug
  Interventions: Drug: Livalo® fixed combination drug

INTERVENTIONS:
Drug: Pitavastatin, Valsartan — Pitavastatin 4mg(2 tablets), Valsartan 160mg(1 tablet)
  Other Names: Livalo, Diovan
  Arms: Pitavastatin + Valsartan
Drug: Livalo® fixed combination drug — Livalo® fixed combination drug(1 tablet)
  Other Names: Livalo, Diovan
  Arms: Livalo fixed combination drug

SUMMARY:
The purpose of this study is to compare pharmacokinetics between Pitavastatin and Valsartan co-administration and Livalo fixed combination drug in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Age 20-55 years at the time of Screening
* BMI 19-26 kg/m2 at the time of Screening

Exclusion Criteria:

* Received other investigational drug within 90 days prior to the first dose of study drug

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-08; Primary Completion 2011-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Cmax of study drugs after single oral administration | 0-48hrs
AUClast of study drugs after single oral administration | 0-48hrs

SECONDARY OUTCOMES:
AUCinf, Tmax and t1/2β of study drugs after single oral administration | 0-48hrs

CONTACTS AND LOCATIONS:
Overall Officials: Kyun Seop Bae, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea